CLINICAL TRIAL: NCT03774251
Title: A Randomized Controlled Trial of Ultrasound-guided Platelet-Rich-Plasma (PRP) Injection Versus Extracorporeal Shock Wave Therapy (ESWT) for Great Trochanter Pain Syndrome (GTPS) With Gluteus Medius or Minimus Tendinopathy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding not secured
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Fredericson, MD, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47910
Record Dates: First submitted 2018-12-04; First posted 2018-12-12 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Greater Trochanter Pain Syndrome, Gluteus Medius Tendinopathy, Gluteus Minimus Tendinopathy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Greater Trochanter Pain Syndrome - PRP Arm (Active Comparator): Individuals with Greater Trochanter Pain Syndrome with MRI evidence of gluteus medius or gluteus minimus tendinopathy, assigned to undergo platelet rich plasma injection
  Interventions: Biological: Platelet-Rich Plasma Injection
- Greater Trochanter Pain Syndrome - ESWT Arm (Active Comparator): Individuals with Greater Trochanter Pain Syndrome with MRI evidence of gluteus medius or gluteus minimus tendinopathy, assigned to extracorporeal shock wave therapy
  Interventions: Device: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Biological: Platelet-Rich Plasma Injection — The patient will undergo a single platelet-rich plasma peritendinous injection
  Arms: Greater Trochanter Pain Syndrome - PRP Arm
Device: Extracorporeal Shock Wave Therapy — The patient will undergo a series of three extracorporeal shock wave therapy treatments to the lateral hip
  Arms: Greater Trochanter Pain Syndrome - ESWT Arm

SUMMARY:
The purpose of this study is to compare the efficacy of ultrasound-guided platelet-rich plasma (PRP) injection versus extracorporeal shock wave therapy for management of refractory Greater Trochanteric Pain Syndrome (GTPS).

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy of ultrasound-guided platelet-rich plasma (PRP) injection versus extracorporeal shock wave therapy for management of refractory Greater Trochanteric Pain Syndrome (GTPS).

GTPS is a common cause of extra-articular lateral hip pain which occurs in up to 10- 25% of the population, and is a common presenting complaint to primary care and Sports Medicine clinics. Previously, most cases of GTPS were diagnosed as trochanteric bursitis, for which the standard treatment focused on relieving inflammation with non-steroidal anti-inflammatory medications and corticosteroid injections. However, corticosteroid injections typically only provide short term pain relief, likely secondary to the fact that the underlying pathology is likely not from an isolated bursal inflammation. Recent studies suggest that in fact the most common cause of GTPS is gluteus medius or minimus tendinopathy or tear. Platelet rich plasma (PRP) has been used in treating tendinopathies and tendon tears throughout the body to promote healing through the concentrated growth factors released from platelets. Extracorporeal shock wave therapy (ESWT) is another treatment which has been used increasingly in the treatment of tendinopathies. The purpose of this randomized prospective study is to compare the efficacy of PRP injection to ESWT in treating patients with a clinical diagnosis of GTPS.

ELIGIBILITY:
Inclusion Criteria:

Individuals with documented diagnosis of greater trochanter pain syndrome, with MRI evidence of gluteus minimus or medius tendinopathy, whose lateral hip pain has been refractory to conservative management with non-steroid anti-inflammatory medications and at least 6 weeks of Physical Therapy.

Exclusion Criteria:

1. Age < 18 or > 65 years
2. Pregnancy
3. Full-thickness tear of the involved gluteal tendons, bursa, and intra-articular structures.
4. Evidence of concomitant injury to the involved lower extremity, including radiculopathy or radiculitis, piriformis syndrome, ischial tuberosity avulsion
5. History of prior steroid injection and Orthobiologic injection or surgery to the involved lower extremity f. Any inflammatory or neoplastic disorder

g. Blood coagulation disorders or use of antiplatelet or anticoagulant drugs h. Severe knee or hip osteoarthritis i. Patients with symptoms of more than 6 months' duration were not considered as patients in the chronic stages of this condition and may require a different therapeutic approach including surgical treatment.

j. Severe Diabetes Mellitus who need insulin injection k. Severe active lumbar radiculopathy with pain, numbness, or weakness in a dermatomal distribution l. Implanted pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pain: VAS | 4 weeks, 3 months, 6 months, 12 months
  Visual Analog Scale (VAS)
Improvement in Function as measured by the International Hip Outcome Tool (iHot) | 4 weeks, 3 months, 6 months, 12 months
Improvement in Function as measured by the Lower extremity functional scale (LEFS) | 4 weeks, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fredericson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine Outpatient Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Wang JH. PRP Treatment Efficacy for Tendinopathy: A Review of Basic Science Studies. Biomed Res Int. 2016;2016:9103792. doi: 10.1155/2016/9103792. Epub 2016 Aug 16. PMID 27610386
- [Background] Rompe JD, Segal NA, Cacchio A, Furia JP, Morral A, Maffulli N. Home training, local corticosteroid injection, or radial shock wave therapy for greater trochanter pain syndrome. Am J Sports Med. 2009 Oct;37(10):1981-90. doi: 10.1177/0363546509334374. Epub 2009 May 13. PMID 19439758
- [Background] Ribeiro AG, Ricioli W Junior, Silva AR, Polesello GC, Guimaraes RP. PRP IN THE TREATMENT OF TROCHANTERIC SYNDROME: A PILOT STUDY. Acta Ortop Bras. 2016 Jul-Aug;24(4):208-212. doi: 10.1590/1413-785220162404159837. PMID 28243176
- [Background] Redmond JM, Chen AW, Domb BG. Greater Trochanteric Pain Syndrome. J Am Acad Orthop Surg. 2016 Apr;24(4):231-40. doi: 10.5435/JAAOS-D-14-00406. PMID 26990713
- [Background] Mani-Babu S, Morrissey D, Waugh C, Screen H, Barton C. The effectiveness of extracorporeal shock wave therapy in lower limb tendinopathy: a systematic review. Am J Sports Med. 2015 Mar;43(3):752-61. doi: 10.1177/0363546514531911. Epub 2014 May 9. PMID 24817008
- [Background] Jacobson JA, Yablon CM, Henning PT, Kazmers IS, Urquhart A, Hallstrom B, Bedi A, Parameswaran A. Greater Trochanteric Pain Syndrome: Percutaneous Tendon Fenestration Versus Platelet-Rich Plasma Injection for Treatment of Gluteal Tendinosis. J Ultrasound Med. 2016 Nov;35(11):2413-2420. doi: 10.7863/ultra.15.11046. Epub 2016 Sep 23. PMID 27663654
- [Background] Seo KH, Lee JY, Yoon K, Do JG, Park HJ, Lee SY, Park YS, Lee YT. Long-term outcome of low-energy extracorporeal shockwave therapy on gluteal tendinopathy documented by magnetic resonance imaging. PLoS One. 2018 Jul 17;13(7):e0197460. doi: 10.1371/journal.pone.0197460. eCollection 2018. PMID 30016333
- [Background] Furia JP, Rompe JD, Maffulli N. Low-energy extracorporeal shock wave therapy as a treatment for greater trochanteric pain syndrome. Am J Sports Med. 2009 Sep;37(9):1806-13. doi: 10.1177/0363546509333014. Epub 2009 May 13. PMID 19439756
- [Background] Fitzpatrick J, Bulsara MK, O'Donnell J, McCrory PR, Zheng MH. The Effectiveness of Platelet-Rich Plasma Injections in Gluteal Tendinopathy: A Randomized, Double-Blind Controlled Trial Comparing a Single Platelet-Rich Plasma Injection With a Single Corticosteroid Injection. Am J Sports Med. 2018 Mar;46(4):933-939. doi: 10.1177/0363546517745525. Epub 2018 Jan 2. PMID 29293361